CLINICAL TRIAL: NCT00180778
Title: Randomised Controlled Trial of Low Dose Steroid +Aspirin +Heparin Versus Aspirin+Heparin Amongst Pregnant Women With APS
Brief Title: Steroids and Antiphospholipid Syndrome- Related Pregnancy Loss
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Literature highlighted unnecessary side effects from the relevant combination.
Sponsor: Imperial College London (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05/Q0403/155; 2005-004182-42
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Steroids

INTERVENTIONS:
Drug: Low dose steroids

SUMMARY:
Does the addition of steroids during the first trimester to the standard aspirin + heparin treatment reduce the miscarriage rates in women with antiphospholipid antibodies and recurrent first trimester miscarriage in those who had an unsuccessful pregnancy with aspirin + heparin?

DETAILED DESCRIPTION:
Over the last decade, the APS has emerged as most important treatable cause of recurrent miscarriages. The pathogenesis of fetal loss in this condition is still remains obscure. Despite the success of aspirin + heparin treatment, some pregnant women with APS repeatedly miscarry even on treatment. The trial is designed to determine if addition of steroids has an success in these women. This is in view of recent in vitro data from our unit reporting that there is an increase decidual cytokine response in APS positive women.

ELIGIBILITY:
Inclusion Criteria:

History of 3 or more consecutive miscarriages and positive antiphospholipid antibodies on at least two occasions more than 6 weeks apart before becoming pregnant and an unsuccessful pregnancy with aspirin + heparin with a karyotype of miscarriage either unavailable or normal (46XX/ 46XY).

Exclusion Criteria:

Abnormal karyotype of women or partner, previous thromboembolism, SLE, diabetes mellitus, hypertension, sensitivity to aspirin, heparin and prednisolone, multiple pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10 (Estimated); Primary Completion 2005-10 (Estimated); Study Completion 2005-10 (Estimated)

PRIMARY OUTCOMES:
Successful pregnancy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Raj Rai, MRCOG, Principal Investigator — Imperial College London
Locations (1):
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837